CLINICAL TRIAL: NCT01186757
Title: A Double Blind (3rd Party Open), Randomized, Placebo Controlled, Dose Escalation Study To Investigate The Safety, Toleration, And Pharmacokinetics Of Multiple Inhaled Doses Of PF-03715455 In Healthy Subjects
Brief Title: Multiple Dose Healthy Volunteer Study of PF-03715455.
Acronym: MD-MULTI DOSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: A9111002
Record Dates: First submitted 2010-08-11; First posted 2010-08-23 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — N-(1-(3-chloro-4-hydroxyphenyl)-3-(1,1-dimethylethyl)-1H-pyrazol-5-yl)-N'-((2-((3-(2-((2-hydroxyethyl)thio)phenyl)-1,2,4-triazolo(4,3-a)pyridin-6-yl)thio)phenyl)methyl)-urea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-03715455 1.6mg BID (Active Comparator)
  Interventions: Drug: PF-03715455
- PF-03715455 4 mg BID (Active Comparator)
  Interventions: Drug: PF-03715455
- PF-03715455 10 mg BID (Active Comparator)
  Interventions: Drug: PF-03715455
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-03715455 — PF-03715455 1.6 mg BID
  Arms: PF-03715455 1.6mg BID
Drug: PF-03715455 — PF-03715455 4mg BID
  Arms: PF-03715455 4 mg BID
Drug: PF-03715455 — PF-03715455 10 mg BID
  Arms: PF-03715455 10 mg BID
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Evaluation of the multiple dose pharmacokinetics of PF-3715455 in healthy volunteers

DETAILED DESCRIPTION:
Healthy volunteer PK study

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Standard healthy volunteer criteria

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single and multiple inhaled doses of PF-03715455, as measured by plasma concentrations - Cmax, Tmax, AUCtau, t½, accumulation ratio (Rac, Rss, Rac,Cmax). | 17 days

SECONDARY OUTCOMES:
Safety and toleration as measured by adverse events, vital signs, 12 lead ECG, blood and urine safety tests and physical examination. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9111002&StudyName=Multiple%20Dose%20Healthy%20Volunteer%20Study%20of%20PF-03715455.